CLINICAL TRIAL: NCT04494425
Title: A Phase 3, Randomized, Multi-center, Open-label Study of Trastuzumab Deruxtecan (T-DXd) Versus Investigator's Choice Chemotherapy in HER2-Low, Hormone Receptor Positive Breast Cancer Patients Whose Disease Has Progressed on Endocrine Therapy in the Metastatic Setting (DESTINY-Breast06)
Brief Title: Study of Trastuzumab Deruxtecan (T-DXd) vs Investigator's Choice Chemotherapy in HER2-low, Hormone Receptor Positive, Metastatic Breast Cancer
Acronym: DB-06
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9670C00001; 2023-505554-18-00 (Registry Identifier: CTIS); 2019-004493-26 (EudraCT Number)
Record Dates: First submitted 2020-07-20; First posted 2020-07-31 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Advanced or Metastatic Breast Cancer
Keywords: Breast Cancer; HR positive; HER2-Low; HER2-Negative; Trastuzumab Deruxtecan (T-DXd; DS-8201a); Anti-HER2-Antibody Drug Conjugate (ADC); DESTINY-Breast06
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; Capecitabine; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Intervention Model Description: The study consists of 2 independent open label treatment arms: trastuzumab deruxtecan and Investigator's choice chemotherapy (paclitaxel, nab-paclitaxel or capecitabine).
Masking Description: This study is an open-label study that will be conducted "Sponsor-blind". To maintain the integrity of the study, Sponsor personnel directly involved in study conduct will not undertake or have access to efficacy data aggregated by treatment group prior to final data readout for the primary endpoint.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trastuzumab deruxtecan (Experimental): Trastuzumab deruxtecan (T-DXd; DS-8201a) arm
  Interventions: Drug: Trastuzumab deruxtecan
- Standard of Care (Active Comparator): Investigator's choice standard of care chemotherapy (capecitabine, paclitaxel, nab-paclitaxel) arm
  Interventions: Drug: Capecitabine; Drug: Paclitaxel; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan by intravenous infusion
  Other Names: DS-8201a; T-DXd
  Arms: Trastuzumab deruxtecan
Drug: Capecitabine — Investigator's choice standard of care single agent chemotherapy; capecitabine tablets will be given orally.
  Arms: Standard of Care
Drug: Paclitaxel — Investigator's choice standard of care single agent chemotherapy; paclitaxel by intravenous infusion.
  Arms: Standard of Care
Drug: Nab-Paclitaxel — Investigator's choice standard of care single agent chemotherapy; nab-paclitaxel by intravenous infusion
  Arms: Standard of Care

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of trastuzumab deruxtecan compared with investigator's choice chemotherapy in human epidermal growth factor receptor (HER)2-low, hormone receptor (HR) positive breast cancer patients whose disease has progressed on endocrine therapy in the metastatic setting.

DETAILED DESCRIPTION:
Eligible patients will be those patients who have had disease progression on at least 2 previous lines of endocrine therapies given for the treatment of metastatic disease or disease progression within 6 months of starting first line treatment for metastatic disease with an endocrine therapy combined with a CDK4/6 inhibitor. All patients must have historically confirmed HR positive (either estrogen receptor and/or progesterone receptor positive), HER2-low (defined as IHC2+/ISH- and IHC 1+) or HER2 IHC >0 <1+ expression, as determined by central laboratory testing results, advanced or metastatic breast cancer.

The study aims to evaluate the efficacy, safety and tolerability of trastuzumab deruxtecan compared with investigator's choice chemotherapy. This study aims to see if trastuzumab deruxtecan allows patients to live longer without the cancer getting worse, or simply to live longer, compared to patients receiving standard of care chemotherapy. This study is also looking to see how the treatment and the cancer affects patients' quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be ≥18 years of age
* Pathologically documented breast cancer that:

  1. is advanced or metastatic
  2. has a history of HER2-low or negative expression by local test, defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested) or HER2 IHC 0 (ISH- or untested)
  3. has HER2-low or HER2 IHC >0 <1+ expression as determined by the central laboratory result established on a tissue sample taken in the metastatic setting
  4. was never previously HER2-positive
  5. is documented HR+ disease in the metastatic setting.
* No prior chemotherapy for advanced or metastatic breast cancer.
* Has adequate tumor samples for assessment of HER2 status
* Must have either:

  1. disease progression within 6 months of starting first line metastatic treatment with an endocrine therapy combined with a CDK4/6 inhibitor or
  2. disease progression on at least 2 previous lines of endocrine therapy with or without a targeted therapy in the metastatic setting. Of note with regards to the ≥2 lines of previous ET requirement: disease recurrence while on the first 24 months of starting adjuvant ET, will be considered a line of therapy; these patients will only require 1 line of ET in the metastatic setting.
* Has protocol-defined adequate organ and bone marrow function

Key Exclusion Criteria:

* Ineligible for all options in the investigator's choice chemotherapy arm
* Lung-specific intercurrent clinically significant illnesses
* Uncontrolled or significant cardiovascular disease or infection
* Prior documented interstitial lung disease (ILD)/ pneumonitis that required steroids, current ILD/ pneumonitis, or suspected ILD/ pneumonitis that cannot be ruled out by imaging at screening.
* Patients with spinal cord compression or clinically active central nervous system metastases
* Prior randomization or treatment in a previous trastuzumab deruxtecan study regardless of treatment arm assignment
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study during the follow up period of a prior interventional study (prescreening for this study while a patient is on treatment in another clinical study is acceptable)

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 866 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2026-06-19 (Estimated)

CONTACTS AND LOCATIONS:
Locations (241):
- United States (26):
  - Research Site, Scottsdale, Arizona
  - Research Site, Springdale, Arkansas
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Lakewood, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Kansas City, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Summit, New Jersey
  - Research Site, Westbury, New York
  - Research Site, Columbus, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
- Argentina (7):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Rosario
- Australia (7):
  - Research Site, Adelaide
  - Research Site, Birtinya
  - Research Site, Darlinghurst
  - Research Site, Murdoch
  - Research Site, South Brisbane
  - Research Site, St Leonards
  - Research Site, Waratah
- Austria (2):
  - Research Site, Graz
  - Research Site, Innsbruck
- Belgium (10):
  - Research Site, Anderlecht
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Namur
  - Research Site, Roeselare
  - Research Site, Sint-Niklaas
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
  - Research Site, Sorocaba
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, CA
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
- China (23):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Dalian
  - Research Site, Foshan
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Copenhagen Ø
  - Research Site, Odense
  - Research Site, Vejle
- France (18):
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Le Mans
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Plerin SUR MER
  - Research Site, Rennes
  - Research Site, Saint-Cloud
  - Research Site, Saint-Herblain
  - Research Site, Tours
  - Research Site, Villejuif
- Germany (7):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Freiburg im Breisgau
  - Research Site, Hanover
  - Research Site, München
  - Research Site, Münster
  - Research Site, Velbert
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
  - Research Site, Szolnok
  - Research Site, Tatabánya
- India (7):
  - Research Site, Bengaluru
  - Research Site, Calicut
  - Research Site, Kolkata
  - Research Site, Marg Jaipur
  - Research Site, New Delhi
  - Research Site, Surat
  - Research Site, Thiruvananthapuram
- Israel (6):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Italy (14):
  - Research Site, Aviano
  - Research Site, Bergamo
  - Research Site, Candiolo
  - Research Site, Cona
  - Research Site, Genova
  - Research Site, Livorno
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Prato
  - Research Site, Tricase, Lecce
  - Research Site, Udine
- Japan (29):
  - Research Site, Akashi-shi
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Hidaka-shi
  - Research Site, Hiroshima
  - Research Site, Isehara
  - Research Site, Kagoshima
  - Research Site, Kashiwa
  - Research Site, Kawasaki-shi
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Naha
  - Research Site, Niigata
  - Research Site, Nishinomiya-shi
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Tsu
  - Research Site, Yokohama
- Mexico (7):
  - Research Site, Alc. Cuauhtémoc
  - Research Site, Guadalajara Jalisco
  - Research Site, Guadalajra
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Nuevo León
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Hengelo
  - Research Site, Leeuwarden
  - Research Site, Rotterdam
  - Research Site, Sittard-Geleen
- Poland (7):
  - Research Site, Bydgoszcz
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Lisbon, Portugal
- Russia (4):
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- Singapore (2):
  - Research Site, Bukit Merah
  - Research Site, Singapore
- South Korea (5):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, El Palmar
  - Research Site, Madrid
  - Research Site, San Sebastián
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Vaxjo
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (8):
  - Research Site, Cambridge
  - Research Site, Cardiff
  - Research Site, Edinburgh
  - Research Site, Guildford
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bardia A, Hu X, Dent R, Yonemori K, Barrios CH, O'Shaughnessy JA, Wildiers H, Pierga JY, Zhang Q, Saura C, Biganzoli L, Sohn J, Im SA, Levy C, Jacot W, Begbie N, Ke J, Patel G, Curigliano G; DESTINY-Breast06 Trial Investigators. Trastuzumab Deruxtecan after Endocrine Therapy in Metastatic Breast Cancer. N Engl J Med. 2024 Dec 5;391(22):2110-2122. doi: 10.1056/NEJMoa2407086. Epub 2024 Sep 15. PMID 39282896
- [Derived] Tarantino P, Tolaney SM, Curigliano G. Trastuzumab deruxtecan (T-DXd) in HER2-low metastatic breast cancer treatment. Ann Oncol. 2023 Oct;34(10):949-950. doi: 10.1016/j.annonc.2023.07.003. Epub 2023 Jul 26. No abstract available. PMID 37499870
- See also: AZ Breast Cancer Study Navigators — http://BreastCancerStudyLocator.com
- See also: Daiichi Sankyo Contact for Clinical Trial Information Phone: 908-992-6400 — http://CTRinfo@dsi.com
- See also: D9670C00001_CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9670C00001&attachmentIdentifier=77d4aa68-56df-404e-80e4-8548804fe415&fileName=D9670C00001_CSP_Redacted.pdf&versionIdentifier=
- See also: D9670C00001_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9670C00001&attachmentIdentifier=da79f59a-5537-4778-857a-106e0db4c436&fileName=D9670C00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: D9670C00001_Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9670C00001&attachmentIdentifier=50fccb14-2a22-4cd5-b60d-b2b25d33ed12&fileName=D9670C00001_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, multi-center, open-label study was conducted in participants with human epidermal growth factor receptor 2 (HER2)-low, hormone receptor-positive (HR+) breast cancer at 273 sites in 28 countries. Results are presented based on primary completion date (PCD) of up to 18 March 2024.
Pre-assignment Details: 866 participants were randomized in a 1:1 ratio to receive trastuzumab deruxtecan (T-DXd) or standard of care: Investigator's choice single agent chemotherapy (capecitabine, paclitaxel or nab-paclitaxel). As pre-specified in the protocol and statistical analysis plan (SAP), results are presented by treatment group.
Groups:
- T-DXd: Participants received T-DXd 5.4 milligram per kilogram (mg/kg) via intravenous (IV) infusion every 3 weeks until disease progression (PD), unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation was met.
- Chemotherapy: Participants received Investigator's choice single-agent chemotherapy (capecitabine 1000 or 1250 mg per meter square [m^2] orally twice daily for 2 weeks followed by a 1-week rest period in 3-week cycles, paclitaxel 80 mg/m^2 via IV infusion every week [qw] in 3-week cycles or nab-paclitaxel 100 mg/m^2 via IV infusion qw for 3 weeks followed by 1-week rest period in 4-week cycles) until PD, unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation was met.
Period: Overall Study
Arm/Group | T-DXd | Chemotherapy
Started (Randomized) | 436 | 430
Randomized and Received Treatment | 434 | 417
Completed | 0 | 0
Not Completed | 436 | 430
Not completed — Death | 160 | 166
Not completed — Withdrawal by Subject | 10 | 40
Not completed — Other | 1 | 1
Not completed — Ongoing at the time of PCD | 265 | 223

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomized participants.
Groups:
- T-DXd: Participants received T-DXd 5.4 mg/kg via IV infusion every 3 weeks until PD, unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation was met.
- Chemotherapy: Participants received Investigator's choice single-agent chemotherapy (capecitabine 1000 or 1250 mg/m^2 orally twice daily for 2 weeks followed by a 1-week rest period in 3-week cycles, paclitaxel 80 mg/m^2 via IV infusion qw in 3-week cycles or nab-paclitaxel 100 mg/m^2 via IV infusion qw for 3 weeks followed by 1-week rest period in 4-week cycles) until PD, unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation was met.
- Total: Total of all reporting groups
Arm/Group | T-DXd | Chemotherapy | Total
Number analyzed (Participants) | 436 | 430 | 866
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (11.46) | 58.2 (10.92) | 58.2 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 436 | 429 | 865
  Male | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 3 | 7
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 154 | 151 | 305
  White | 231 | 230 | 461
  Other | 7 | 12 | 19
  Not reported | 39 | 34 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 32 | 60
  Not Hispanic or Latino | 397 | 387 | 784
  Missing | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Assessed by Blinded Independent Central Review (BICR) in the Hormone Receptor-Positive (HR+), Human Epidermal Growth Factor Receptor 2 (HER2)-Low Population
Description: PFS per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) assessed by BICR was defined as the time from the date of randomization until the date of PD, as defined or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anticancer therapy prior to progression. PD was defined as at least a 20% increase in the sum of diameters of target lesions (TLs), taking as reference the smallest previous sum of diameters (nadir), this included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 millimeter (mm) from nadir. Median PFS was calculated using Kaplan-Meier method and its confidence interval (CI) using Brookmeyer-Crowley method.
Time Frame: Response evaluations performed at screening, every 6 weeks (q6w) ± 1 week from randomization for 48 weeks, and then every 9 weeks (q9w) ± 1 week, starting at Week 48 until PD, up to PCD of 18 March 2024 (maximum of approximately 43.85 months)
Population: The HER2-low population included the subset of participants in the ITT population with HER2 immunohistochemistry (IHC) 2+/ in situ hybridization (ISH)- and IHC 1+ as determined per the interactive response technology (IRT) data for HER2 IHC expression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 359 | 354
months | 13.2 [11.4 to 15.2] | 8.1 [7.0 to 9.0]
Statistical Analysis 1: Comparison: T-DXd vs Chemotherapy; Test type: Superiority; p < 0.0001, Log Rank; The analysis was performed using the stratified log-rank test; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.52 to 0.75] — HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for prior cyclin-dependent kinase (CDK)4/6 inhibitor use (yes versus no) and HER2 IHC expression (IHC 1+ versus IHC 2+/ISH-) and ties handled by Efron approach

2. Secondary Outcome: Overall Survival (OS) in the Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-low Population
Description: OS was defined as the time from the date of randomization until death due to any cause regardless of whether the participant withdrew from randomized therapy or received another anticancer therapy. Median OS was calculated using Kaplan-Meier method and its CI using Brookmeyer-Crowley method.
Time Frame: From date of randomization until death due to any cause, up to PCD of 18 March 2024 (maximum of approximately 43.85 months)
Population: The HER2-low population included the subset of participants in the ITT population with HER2 IHC 2+/ISH- and IHC 1+ as determined per the IRT data for HER2 IHC expression.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 359 | 354
months | 28.9 [25.7 to 33.7] | 27.1 [23.5 to 29.9]

3. Secondary Outcome: Progression-Free Survival Assessed by Blinded Independent Central Review in the Intent-to-Treat, Human Epidermal Growth Factor Receptor 2 Immunohistochemistry (IHC) >0 <1+ and Human Epidermal Growth Factor Receptor 2-low Population
Description: PFS per RECIST 1.1 assessed by BICR was defined as the time from the date of randomization until the date of PD, as defined or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anticancer therapy prior to progression. PD was defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir), this included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 mm from nadir. Median PFS was calculated using Kaplan-Meier method and its CI using Brookmeyer-Crowley method.
Time Frame: Response evaluations performed at screening, q6w ± 1 week from randomization for 48 weeks, and then q9w ± 1 week, starting at Week 48 until PD, up to PCD of 18 March 2024 (maximum of approximately 43.85 months)
Population: ITT population: all randomized participants. HER2 IHC >0 <1+ population: subset of participants included in ITT population with HER2 IHC >0 <1+ as determined by central laboratory testing and who have had at least 24 weeks of follow-up at time of interim futility PCD. HER2-low population: subset of participants in ITT population with HER2 IHC 2+/ISH- and IHC 1+ as determined per IRT data for HER2 IHC expression. Only participants with data collected in specified categories are reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 436 | 430
months
  ITT Population | 13.2 [12.0 to 15.2] | 8.1 [7.0 to 9.0]
  HER2 IHC >0 <1+ Population: number analyzed (Participants) | 76 | 76
  HER2 IHC >0 <1+ Population | 13.2 [9.8 to 17.3] | 8.3 [5.8 to 15.2]
  HER2-low Population: number analyzed (Participants) | 359 | 354
  HER2-low Population | 12.8 [11.1 to 13.2] | 7.0 [6.4 to 7.5]

4. Secondary Outcome: Overall Survival (OS) in the Intent-to-Treat Population
Description: as for outcome 2
Time Frame: as for outcome 2
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 436 | 430
months | 28.9 [26.4 to 32.7] | 27.4 [23.9 to 29.9]

5. Secondary Outcome: Progression-Free Survival Assessed by Investigator in the Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-low Population
Description: PFS per RECIST 1.1 assessed by Investigator was defined as the time from the date of randomization until the date of PD, as defined or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anticancer therapy prior to progression. PD was defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir), this included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 mm from nadir. Median PFS was calculated using Kaplan-Meier method and its CI using Brookmeyer-Crowley method.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 359 | 354
months | 12.8 [11.1 to 13.2] | 7.0 [6.4 to 7.5]

6. Secondary Outcome: Objective Response Rate (ORR) Assessed by Blinded Independent Central Review and Investigator in the Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-low Population
Description: ORR per RECIST 1.1 assessed by BICR and Investigator was defined as the percentage of participants with at least 1 visit response of complete response (CR) or partial response (PR). CR was defined as disappearance of all TLs since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm. PR was defined as at least a 30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 359 | 354
percentage of participants
  BICR Assessment | 60.4 | 37.9
  Investigator Assessment | 60.4 | 40.4

7. Secondary Outcome: Duration of Response (DOR) Assessed by Blinded Independent Central Review and Investigator in the Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-low Population
Description: DOR per RECIST v1.1 was defined as the time from the date of first documented response until date of documented progression or death in the absence of PD. PD was defined as at least a 20% increase in the sum of diameters of TLs, taking as reference the smallest previous sum of diameters (nadir), this included the baseline sum if that was the smallest on study. In addition to the relative increase of 20%, the sum must demonstrate an absolute increase of at least 5 mm from nadir. Median DOR was calculated using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: The HER2-low population included the subset of participants in the ITT population with HER2 IHC 2+/ISH- and IHC 1+ as determined per the IRT data for HER2 IHC expression. Only participants with response in each specified category are reported.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 217 | 143
months
  BICR Assessment: number analyzed (Participants) | 217 | 134
  BICR Assessment | 13.6 [6.2 to 24.9] | 7.3 [4.2 to 15.2]
  Investigator Assessment | 12.0 [6.6 to 20.0] | 6.9 [3.1 to 11.1]

8. Secondary Outcome: Objective Response Rate Assessed by Blinded Independent Central Review and Investigator in the Intent-to-Treat and Human Epidermal Growth Factor Receptor 2 Immunohistochemistry >0 <1+ Population
Description: ORR per RECIST 1.1 assessed by BICR and Investigator was defined as the percentage of participants with at least 1 visit response of CR or PR. CR was defined as disappearance of all TLs since baseline. Any pathological lymph nodes selected as TLs must have a reduction in short axis diameter to <10 mm. PR was defined as at least a 30% decrease in the sum of the diameters of TL, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 3
Population: The ITT population included all randomized participants. The HER2 IHC >0 <1+ population included subset of participants included in ITT population with HER2 IHC >0 <1+ as determined by central laboratory testing and who have had at least 24 weeks of follow-up at time of interim futility PCD. Only participants with data collected in specified categories are reported.
Measure: Number; unit: percentage of participants
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 436 | 430
percentage of participants
  BICR Assessment: ITT Population | 61.5 | 36.7
  Investigator Assessment: ITT Population | 61.5 | 38.8
  BICR Assessment: HER2 IHC >0 <1+ Population: number analyzed (Participants) | 76 | 76
  BICR Assessment: HER2 IHC >0 <1+ Population | 67.1 | 31.6
  Investigator Assessment: HER2 IHC >0 <1+ Population: number analyzed (Participants) | 76 | 76
  Investigator Assessment: HER2 IHC >0 <1+ Population | 65.8 | 31.6

9. Secondary Outcome: Duration of Response Assessed by Blinded Independent Central Review and Investigator in the Intent-to-Treat Population
Description: as for outcome 7
Time Frame: as for outcome 3
Population: The ITT population included all randomized participants. Only participants with response in each specified category are reported.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 268 | 167
months
  BICR Assessment: number analyzed (Participants) | 268 | 158
  BICR Assessment | 13.7 [6.5 to 24.9] | 7.3 [4.2 to 15.9]
  Investigator Assessment | 12.1 [6.8 to 20.0] | 6.9 [3.0 to 12.5]

10. Secondary Outcome: Time From Randomization to Second Progression or Death (PFS2) in the Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-low and Intent-to-Treat Population
Description: PFS2 was defined as time from randomization to second progression (the earliest of the progression event subsequent to first subsequent therapy) or death; second progression was defined according to local standard clinical practice and might involve any of the following: objective radiological imaging, symptomatic progression, or death. Median PFS2 was calculated using Kaplan-Meier method and its CI using Brookmeyer-Crowley method.
Time Frame: as for outcome 3
Population: The HER2-low population included subset of participants in ITT population with HER2 IHC 2+/ISH- and IHC 1+ as determined per IRT data for HER2 IHC expression. The ITT population included all randomized participants. Only participants with data collected in specified categories are reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 436 | 430
months
  HER2-low Population: number analyzed (Participants) | 359 | 354
  HER2-low Population | 20.0 [18.9 to 23.8] | 14.5 [12.9 to 15.5]
  ITT Population | 20.3 [18.9 to 23.8] | 14.7 [13.5 to 15.9]

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant administered a medicinal product and which did not necessarily had a causal relationship with this treatment. A serious adverse event (SAE) was an AE occurring during any study phase, that fulfilled 1 or more of following criteria: resulted in death, was immediately life-threatening, required in-participant hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability or incapacity, was congenital abnormality or birth defect, and was an important medical event that jeopardized participant or required medical treatment to prevent 1 of outcomes listed above. TEAE was any AE that occurred, having been absent before the first dose of study drug, or had worsened in severity or seriousness after initiation of the study drug until the 40-day (+7 days) safety follow-up visit.
Time Frame: From first dose of study drug (Day 1) up to PCD of 18 March 2024 (maximum of approximately 43.85 months)
Population: The Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 434 | 417
Participants
  TEAEs | 429 | 397
  TESAEs | 88 | 67

12. Secondary Outcome: Serum Concentration of Trastuzumab Deruxtecan (T-DXd), Total Anti-Human Epidermal Growth Factor Receptor 2 Antibody and MAAA-1181a
Description: Blood samples were collected at indicated time points to determine the concentration of T-DXd, total anti-HER2 antibody and MAAA-1181a in serum.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 4, 6 and 8; 15 minutes post-dose on Day 1 of Cycles 1, 2 and 4; and 5 hours post-dose on Day 1 of Cycle 1 (each cycle is 21 days)
Population: The Pharmacokinetic population included all participants who received at least 1 dose of T-DXd per the protocol for whom any post-dose data were available. Only participants with data collected in specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | T-DXd
Number analyzed (Participants) | 407
micrograms per milliliter (mcg/mL)
  T-DXd: Day 1: pre-dose, Cycle 1: number analyzed (Participants) | 5
  T-DXd: Day 1: pre-dose, Cycle 1 | NA (NA) — NA indicated that mean and standard deviation (SD) were not estimable as the values were below the lower limit of quantification (LLOQ). LLOQ was 0.4 mcg/mL.
  T-DXd: Day 1: pre-dose, Cycle 2: number analyzed (Participants) | 402
  T-DXd: Day 1: pre-dose, Cycle 2 | 4.35225 (8.958729)
  T-DXd: Day 1: pre-dose, Cycle 4: number analyzed (Participants) | 374
  T-DXd: Day 1: pre-dose, Cycle 4 | 8.21037 (9.464435)
  T-DXd: Day 1: pre-dose, Cycle 6: number analyzed (Participants) | 336
  T-DXd: Day 1: pre-dose, Cycle 6 | 8.65950 (4.753592)
  T-DXd: Day 1: pre-dose, Cycle 8: number analyzed (Participants) | 304
  T-DXd: Day 1: pre-dose, Cycle 8 | 11.31496 (22.894112)
  T-DXd: Day 1: 15 minutes post-dose, Cycle 1: number analyzed (Participants) | 367
  T-DXd: Day 1: 15 minutes post-dose, Cycle 1 | 135.90160 (102.989325)
  T-DXd: Day 1: 15 minutes post-dose, Cycle 2: number analyzed (Participants) | 378
  T-DXd: Day 1: 15 minutes post-dose, Cycle 2 | 136.74872 (108.860006)
  T-DXd: Day 1: 15 minutes post-dose, Cycle 4: number analyzed (Participants) | 347
  T-DXd: Day 1: 15 minutes post-dose, Cycle 4 | 124.60481 (39.812165)
  T-DXd: Day 1: 5 hours post-dose, Cycle 1: number analyzed (Participants) | 366
  T-DXd: Day 1: 5 hours post-dose, Cycle 1 | 123.82288 (30.513998)
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 1: number analyzed (Participants) | 3
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 1 | NA (NA) — NA indicated that mean and SD were not estimable as the values were below the LLOQ. LLOQ was 0.4 mcg/mL.
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 2: number analyzed (Participants) | 390
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 2 | 5.75841 (11.351915)
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 4: number analyzed (Participants) | 370
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 4 | 12.00513 (11.087226)
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 6: number analyzed (Participants) | 333
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 6 | 13.97891 (8.720790)
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 8: number analyzed (Participants) | 302
  Total anti-HER2 antibody: Day 1: pre-dose, Cycle 8 | 17.47641 (27.144299)
  Total anti-HER2 antibody: Day 1: 15 minutes post-dose, Cycle 1: number analyzed (Participants) | 367
  Total anti-HER2 antibody: Day 1: 15 minutes post-dose, Cycle 1 | 141.27586 (114.137606)
  Total anti-HER2 antibody: Day 1: 15 minutes post-dose, Cycle 2: number analyzed (Participants) | 377
  Total anti-HER2 antibody: Day 1: 15 minutes post-dose, Cycle 2 | 146.17993 (134.780719)
  Total anti-HER2 antibody: Day 1: 15 minutes post-dose, Cycle 4: number analyzed (Participants) | 345
  Total anti-HER2 antibody: Day 1: 15 minutes post-dose, Cycle 4 | 131.06830 (44.228380)
  Total anti-HER2 antibody: Day 1: 5 hours post-dose, Cycle 1: number analyzed (Participants) | 363
  Total anti-HER2 antibody: Day 1: 5 hours post-dose, Cycle 1 | 119.64619 (26.591288)
  MAAA-1181a: Day 1: pre-dose, Cycle 1: number analyzed (Participants) | 3
  MAAA-1181a: Day 1: pre-dose, Cycle 1 | NA (NA) — NA indicated that mean and SD were not estimable as the values were below the LLOQ. LLOQ was 0.00001 mcg/mL.
  MAAA-1181a: Day 1: pre-dose, Cycle 2 | 0.261850 (0.2096642)
  MAAA-1181a: Day 1: pre-dose, Cycle 4: number analyzed (Participants) | 380
  MAAA-1181a: Day 1: pre-dose, Cycle 4 | 0.401004 (0.2825761)
  MAAA-1181a: Day 1: pre-dose, Cycle 6: number analyzed (Participants) | 336
  MAAA-1181a: Day 1: pre-dose, Cycle 6 | 0.446237 (0.2957478)
  MAAA-1181a: Day 1: pre-dose, Cycle 8: number analyzed (Participants) | 307
  MAAA-1181a: Day 1: pre-dose, Cycle 8 | 0.432894 (0.2819292)
  MAAA-1181a: Day 1: 15 minutes post-dose, Cycle 1: number analyzed (Participants) | 367
  MAAA-1181a: Day 1: 15 minutes post-dose, Cycle 1 | 6.014366 (3.1859583)
  MAAA-1181a: Day 1: 15 minutes post-dose, Cycle 2: number analyzed (Participants) | 376
  MAAA-1181a: Day 1: 15 minutes post-dose, Cycle 2 | 2.985606 (1.9276120)
  MAAA-1181a: Day 1: 15 minutes post-dose, Cycle 4: number analyzed (Participants) | 348
  MAAA-1181a: Day 1: 15 minutes post-dose, Cycle 4 | 2.411409 (1.5862547)
  MAAA-1181a: Day 1: 5 hours post-dose, Cycle 1: number analyzed (Participants) | 363
  MAAA-1181a: Day 1: 5 hours post-dose, Cycle 1 | 13.917874 (6.5178612)

13. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Scale Score at Week 91
Description: EORTC QLQ-C30 is a 30-item self-administered questionnaire grouped into 5 multi-item functional scales(physical,role,emotional,cognitive and social),3 multiitem symptom scales(fatigue,pain and nausea/vomiting),2-item global QoL scale,5 single items assessing additional symptoms reported by cancer participants(dyspnea,loss of appetite,insomnia,constipation and diarrhea). All but 2 questions have 4-point scales:1:not at all,2:a little,3:quite a bit,4:very much.2 questions concerning global health status and QoL have 7-point scales with responses ranging from 1:very poor to 7:excellent;higher score:better level of functioning/greater degree of symptoms.For each of 15 scales,final scores were averaged from scores of component items,transformed,range: 0 to 100;higher scores:better functioning,better health related (HR)QoL,or greater level of symptoms(higher scores:opposite interpretations for functioning/QoL and symptoms/problems).Baseline:last observed measurement prior to randomization.
Time Frame: Baseline (Day 1) and Week 91
Population: The ITT population included all randomized participants. Only participants with data collected in specified categories are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 44 | 22
score on a scale
  Physical Functioning | -7.88 (17.389) | -4.85 (13.520)
  Role Functioning | -14.77 (21.631) | -12.12 (26.318)
  Emotional Functioning | -6.06 (25.440) | 1.52 (22.218)
  Cognitive Functioning | -8.71 (22.872) | -6.82 (19.009)
  Social Functioning | -10.98 (23.000) | -7.58 (21.656)
  Fatigue | 11.87 (24.367) | 8.59 (18.444)
  Pain | -1.89 (21.025) | -0.76 (24.922)
  Nausea/Vomiting | 9.85 (19.128) | -0.76 (12.037)
  Global Health Status/QoL | -7.77 (23.529) | -10.61 (22.150)
  Dyspnea | 6.06 (23.041) | 1.52 (21.767)
  Loss of Appetite | 12.88 (30.682) | 6.06 (19.616)
  Insomnia | 6.06 (26.190) | -15.15 (24.618)
  Constipation | 11.36 (30.452) | 1.52 (12.503)
  Diarrhea | 6.82 (19.792) | 13.64 (28.469)

14. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Breast Module 45 (BR45) Scale Score at Week 58
Description: EORTC QLQ-BR45 is an updated version of the BR23. Self-administered instrument includes original 23-items yielding 5 multi-item scores (body image, sexual functioning, arm symptoms, breast symptoms, and systemic therapy side effects). Additional 22 items yield 4 additional multi-item scales (breast satisfaction, endocrine therapy symptoms, skin mucosis symptoms, and endocrine sexual symptoms). Single items assess sexual enjoyment, future perspective and being upset by hair loss. Items are scored on a 4-point verbal rating scale: 1: not at all, 2: a little, 3: quite a bit, and 4: very much; higher score: better level of functioning or greater degree of symptoms. Scores of these scales were averaged from scores of component items, transformed, and ranged from 0 to 100; higher scores for functioning scales or items indicate better functioning, whereas higher scores for symptom scales or items represent a higher level of symptoms. Baseline:last observed measurement prior to randomization.
Time Frame: Baseline (Day 1) and Week 58
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 107 | 80
score on a scale
  Body Image | -3.12 (23.585) | -5.42 (22.349)
  Sexual Functioning | -2.96 (12.708) | 1.46 (14.081)
  Arm Symptoms | -5.30 (20.496) | -3.06 (18.540)
  Breast Symptoms | -2.41 (17.132) | -2.19 (12.631)
  Systemic Therapy Side Effects | 5.65 (15.536) | 3.99 (15.536)
  Breast Satisfaction: number analyzed (Participants) | 107 | 78
  Breast Satisfaction | 2.65 (30.982) | 0.85 (31.428)
  Endocrine Therapy Symptoms | -0.14 (11.316) | 0.17 (12.458)
  Skin Mucosis Symptoms | 4.67 (14.721) | 12.22 (18.232)
  Endocrine Sexual Symptoms: number analyzed (Participants) | 107 | 79
  Endocrine Sexual Symptoms | 3.66 (20.831) | 2.00 (15.969)
  Sexual Enjoyment: number analyzed (Participants) | 11 | 12
  Sexual Enjoyment | -3.03 (17.979) | 0.00 (20.101)
  Future Perspective | 8.72 (32.161) | 11.25 (29.022)
  Being Upset By Hair Loss: number analyzed (Participants) | 27 | 9
  Being Upset By Hair Loss | 2.47 (34.500) | 0.00 (40.825)

15. Secondary Outcome: Time to Deterioration in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 Scale Score
Description: Time to deterioration was defined as the time from randomization until the date of the first clinically meaningful deterioration that was confirmed at next available assessment, at least 14 days apart, regardless of whether the participant withdrew from study treatment or receives another anti-cancer therapy prior to deterioration.
Time Frame: From randomization until date of first symptom deterioration that is confirmed, up to PCD of 18 March 2024 (maximum of approximately 43.85 months)
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T-DXd | Chemotherapy
Number analyzed (Participants) | 436 | 430
months
  Physical Functioning | 18.0 [15.9 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 9.9 [6.9 to 15.2]
  Role Functioning | 10.3 [6.9 to 14.6] | 5.5 [4.1 to 6.9]
  Emotional Functioning | 28.2 [18.6 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 17.3 [12.4 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  Cognitive Functioning | 11.8 [8.3 to 16.6] | 9.9 [7.8 to 13.8]
  Social Functioning | 11.7 [7.6 to 16.3] | 7.7 [6.2 to 10.4]
  Fatigue | 4.3 [3.4 to 7.7] | 2.9 [2.2 to 4.2]
  Pain | 22.0 [17.2 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 6.3 [4.8 to 9.6]
  Nausea/Vomiting | 3.5 [2.8 to 5.6] | 13.8 [7.7 to 21.5]
  Global Health Status/QoL | 11.3 [8.3 to 14.7] | 10.5 [7.7 to 13.3]
  Dyspnea | 20.0 [19.3 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 20.8 [13.1 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  Loss of Appetite | 8.3 [5.0 to 11.7] | 13.8 [9.6 to 16.1]
  Insomnia | NA [17.3 to NA] — NA indicated that the median and upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 15.2 [12.4 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  Constipation | 9.2 [5.5 to 12.5] | 22.0 [15.9 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  Diarrhea | 29.0 [17.2 to NA] — NA indicated that the upper limit of 95% CI was not estimable due to insufficient number of participants with events. | 16.5 [13.9 to 23.4]

16. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) Against Trastuzumab Deruxtecan
Description: Blood samples were collected at indicated timepoints to determine ADA. Treatment-induced ADA was defined as ADA positive post-baseline and not detected at baseline (negative or missing). Treatment-boosted ADA was defined as a baseline positive ADA titer that was boosted to a 4-fold or higher-level following drug administration.
Time Frame: From Day 1 up to PCD of 18 March 2024 (maximum of approximately 43.85 months)
Population: The ADA population included all participants who received at least 1 dose of T-DXd and who had a non-missing ADA result at any time.
Measure: Count of Participants; unit: Participants
Arm/Group | T-DXd
Number analyzed (Participants) | 433
Participants
  Treatment-induced ADA | 22
  Treatment-boosted ADA | 0

17. Secondary Outcome: Time to First Subsequent Treatment or Death (TFST) in the Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-low and Intent-to-Treat Population
Description: TFST was defined as time from randomization to the start date of the first subsequent anti-cancer therapy after discontinuation of randomized treatment or death due to any cause.
Time Frame: From Day 1 up to 64 months
Reporting Status: Not Posted, anticipated posting 2025-12

18. Secondary Outcome: Time to Second Subsequent Treatment or Death (TSST) in the Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-low and Intent-to-Treat Population
Description: TSST was defined as time from randomization to the start date of the second subsequent anti-cancer therapy after discontinuation of randomized treatment or death due to any cause.
Time Frame: From Day 1 up to 64 months
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to PCD of 18 March 2024 (maximum of approximately 43.85 months).
Description: The Safety population included all participants who received at least 1 dose of study drug. All-cause mortality was reported in ITT population.
Arm/Group | T-DXd | Chemotherapy
All-Cause Mortality (participants affected / at risk) | 161/436 | 174/430
Serious Adverse Events (participants affected / at risk) | 88/434 | 67/417
Other Adverse Events (participants affected / at risk) | 427/434 | 383/417
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DXd (N=434) | Chemotherapy (N=417)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Femoral hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
General physical health deterioration (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 7 (7) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 5 (5)
Cytomegalovirus hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Human ehrlichiosis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Meningoencephalitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Proteus infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DXd (N=434) | Chemotherapy (N=417)
Abdominal pain (Gastrointestinal disorders) | 45 (61) | 34 (36)
Abdominal pain upper (Gastrointestinal disorders) | 35 (57) | 20 (21)
Neutropenia (Blood and lymphatic system disorders) | 76 (199) | 63 (148)
Constipation (Gastrointestinal disorders) | 136 (179) | 60 (79)
Diarrhoea (Gastrointestinal disorders) | 148 (228) | 112 (177)
Dry mouth (Gastrointestinal disorders) | 24 (24) | 16 (16)
Dyspepsia (Gastrointestinal disorders) | 50 (63) | 20 (23)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (33) | 7 (7)
Nausea (Gastrointestinal disorders) | 301 (585) | 126 (198)
Stomatitis (Gastrointestinal disorders) | 57 (75) | 37 (45)
Vomiting (Gastrointestinal disorders) | 145 (286) | 48 (63)
Asthenia (General disorders) | 98 (182) | 71 (102)
Anaemia (Blood and lymphatic system disorders) | 157 (288) | 106 (216)
Fatigue (General disorders) | 117 (156) | 83 (95)
Malaise (General disorders) | 35 (54) | 18 (23)
Oedema peripheral (General disorders) | 36 (39) | 59 (67)
Pyrexia (General disorders) | 52 (64) | 28 (35)
COVID-19 (Infections and infestations) | 101 (107) | 51 (53)
Nasopharyngitis (Infections and infestations) | 24 (27) | 15 (19)
Urinary tract infection (Infections and infestations) | 28 (40) | 20 (23)
Alanine aminotransferase increased (Investigations) | 93 (142) | 48 (85)
Aspartate aminotransferase increased (Investigations) | 117 (190) | 44 (80)
Blood alkaline phosphatase increased (Investigations) | 48 (62) | 17 (26)
Blood bilirubin increased (Investigations) | 29 (48) | 20 (42)
Ejection fraction decreased (Investigations) | 35 (41) | 12 (13)
Gamma-glutamyltransferase increased (Investigations) | 40 (46) | 9 (13)
Lymphocyte count decreased (Investigations) | 27 (69) | 11 (30)
Neutrophil count decreased (Investigations) | 99 (433) | 66 (265)
Platelet count decreased (Investigations) | 60 (160) | 15 (40)
Weight decreased (Investigations) | 32 (35) | 8 (9)
White blood cell count decreased (Investigations) | 79 (376) | 53 (265)
Decreased appetite (Metabolism and nutrition disorders) | 112 (183) | 47 (53)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25 (48) | 12 (25)
Hypokalaemia (Metabolism and nutrition disorders) | 52 (87) | 14 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 (38) | 45 (53)
Back pain (Musculoskeletal and connective tissue disorders) | 36 (40) | 34 (37)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (25) | 27 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (30) | 23 (27)
Dizziness (Nervous system disorders) | 37 (45) | 26 (26)
Dysgeusia (Nervous system disorders) | 51 (55) | 24 (24)
Headache (Nervous system disorders) | 74 (111) | 42 (44)
Neuropathy peripheral (Nervous system disorders) | 8 (11) | 36 (39)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (13) | 49 (57)
Insomnia (Psychiatric disorders) | 32 (34) | 19 (19)
Dry eye (Eye disorders) | 28 (30) | 18 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 69 (84) | 38 (47)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (30) | 41 (42)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 44 (56) | 15 (16)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 22 (26) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 210 (212) | 87 (89)
Dry skin (Skin and subcutaneous tissue disorders) | 22 (24) | 15 (15)
Leukopenia (Blood and lymphatic system disorders) | 30 (66) | 17 (34)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4) | 145 (176)
Rash (Skin and subcutaneous tissue disorders) | 26 (30) | 31 (35)
Hypertension (Vascular disorders) | 27 (36) | 23 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT04494425/Prot_002.pdf
  • Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT04494425/SAP_003.pdf